CLINICAL TRIAL: NCT05134675
Title: Does Homebrewing Beer Affect Urinary Tract Symptoms and Bladder Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Kaan Yildiz, Principal Investigator, Ankara Training and Research Hospital
Other Study IDs: CB2021
Record Dates: First submitted 2021-11-15; First posted 2021-11-26 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Addiction, Alcohol; Urinary Tract Disease
Keywords: beer; urinary tract
MeSH Terms: conditions — Alcoholism; Urologic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Consumption: Patients consuming homemade beer
  Interventions: Dietary Supplement: Homemade beer
- Not consumption: Patients are not consuming homemade beer
  Interventions: Dietary Supplement: Homemade beer

INTERVENTIONS:
Dietary Supplement: Homemade beer — The data of patients who consume and do not consume homemade beer will be cross-sectionally evaluated and compared.
  Other Names: Homebrewing beer

SUMMARY:
In this study, investigators aim to reveal the harmful effects of increasing consumption of homemade beer in recent years on the urinary tract. The high amount of carbonyl compounds in the content of homemade beer has been proven by studies. In this study, which will be conducted in the form of a questionnaire, it is aimed to evaluate the effects of the consumption of homemade beer and the long-term exposure of the urinary system to carbonyl compounds.

DETAILED DESCRIPTION:
Homemade and craft beers are perceived as a popular alternative to beers produced on a larger scale in recent years, due to the choice of consumers according to different taste preferences and the raw materials used for brewing. According to nationally representative survey data from the American Homebrewers Association (AHA), the U.S. had an estimated 1.1 million homebrew brewers in 2017, with annual homebrew beer production in excess of 1.4 million barrels (about 1% of annual U.S. beer production). Again in 2017, 40% of home brewers started production within the last 4 years. Due to the prohibitions that have arisen due to the pandemic all over the world, the production of homemade beer has reached its peak today. In recent years, home-made beer consumption has gained popularity in parallel with low-alcohol and non-alcoholic beers, which are prone to microbial spoilage, due to the ease of access to the material, financial returns and hobby acquisition.

Homemade beer is typically more susceptible to spoilage as it is not pasteurized or sterile filtered. The microbiota, which is associated with organic raw materials, fruits, herbs, honey, spices and vegetables, and non-traditional starch-rich ingredients added to produce different aromas and flavors, increases the risk of spoilage. In addition, home brewers often lack the advantages of a sophisticated microbiological laboratory, and optimal temperature control during brewing and storage cannot be guaranteed. In addition to the fermentation conditions (time and temperature), yeast strain and mash composition (types of grain used in malting, mashing/boiling conditions) can also affect the chemical profile of beer, resulting in a wide variety of components. Carbonyl compounds [acetaldehyde, acrolein, ethyl carbamate (EC) and formaldehyde] are particularly toxic compounds that can occur. Acetaldehyde, acrolein, and formaldehyde are highly reactive due to their electrophilic nature, so they easily react with biological nucleophilic targets such as proteins, RNA, and DNA.

ELIGIBILITY:
Inclusion Criteria:

* Homemade beer consumption and not consumption

Exclusion Criteria

* Bleeding disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who consume and do not consume homemade beer will be included in our study. Homemade beer consumption definition, for more than 3 months; regular consumption of 1 or more home-made beer in 1 week for women was considered as 2 or more home-made beer consumption in 1 week for men.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-06-16 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Rates of urinary tract symptoms | 3 months
  Rates of urinary tract symptoms who consumed the homemade beer
Rates of bladder cancer | 3 months
  Rates of bladder cancer who consumed the homemade beer

CONTACTS AND LOCATIONS:
Overall Officials: Ali Kaan Yildiz, Principal Investigator — Ankara Training and Resarch Hospital
Locations (1):
- Ankara Training and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lachenmeier DW, Przybylski MC, Rehm J. Comparative risk assessment of carcinogens in alcoholic beverages using the margin of exposure approach. Int J Cancer. 2012 Sep 15;131(6):E995-1003. doi: 10.1002/ijc.27553. Epub 2012 Apr 17. PMID 22447328